CLINICAL TRIAL: NCT04984863
Title: Clinical Usefulness of Magnetically Controlled Capsule Endoscopy in Assessing Efficacy of Gastro-oesophageal Varices in Patients With Liver Cirrhosis Treated Under Gastroscopy: a Prospective, Multicenter Trial
Brief Title: MCCE in Assessing Efficacy of Gastro-oesophageal Varices
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RuijinH20190228
Record Dates: First submitted 2021-01-31; First posted 2021-08-02 (Actual); Last update posted 2021-08-02 (Actual); Status verified 2021-01

CONDITIONS: Gastroesophageal Varices
MeSH Terms: interventions — Endoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- magnetically controlled capsule endoscopy (Experimental): magnetically controlled capsule endoscopy to evaluate the efficacy of the treatment of gastroesophageal varices
  Interventions: Device: Magnetically controlled capsule endoscopy

INTERVENTIONS:
Device: Magnetically controlled capsule endoscopy — Magnetically controlled capsule endoscopy (MCE) is a non-invasive detection method independently developed in China that covers the whole digestive tract (except colon) mucosa.

SUMMARY:
This study proposed for the first time the use of MCE to evaluate the efficacy of the treatment of gastroesophageal varices, and compared the examination results with the gold standard to explore whether MCE could replace the electronic gastroscopy as the preferred non-invasive evaluation method for the treatment of gastroesophageal varices.

DETAILED DESCRIPTION:
Gastro-esophageal varices is one of the complications of portal hypertension in cirrhosis. For patients with moderate to severe varicose veins, international guidelines recommend active treatment, including endoscopic therapy such as endoscopic band ligation (EBL) and interventional radiotherapy such as balloon-occluded retrograde transvenous obliteration (B-RTO)Electronic gastroscopy is the gold standard for the diagnosis of varicose veins at higher blood risk (varicose veins requiring retreatment). However, it is relatively invasive and uncomfortable in the examination process, so that patients with gain-and-compensation cirrhosis are often unwilling to accept it, which is not conducive to the standardized follow-up after the treatment of gastro-esophageal varices.Magnetically controlled capsule endoscopy (MCE) is a non-invasive detection method independently developed in China that covers the whole digestive tract (except colon) mucosa. Patients only need to swallow a capsule endoscope to make repeated observation for many times, and the examination process is painless. It is an ideal method for diagnosing varicose veins with high blood risk (varicose veins that need treatment). Therefore, this study proposed for the first time the use of MCE to evaluate the efficacy of the treatment of gastroesophageal varices, and compared the examination results with the gold standard to explore whether MCE could replace the electronic gastroscopy as the preferred non-invasive evaluation method for the treatment of gastroesophageal varices.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* Confirmed cirrhosis by clinical or pathological biopsy
* Previous endoscopic treatment of esophageal and gastric varices, including but not limited to sclerotherapy, injection of tissue adhesives, skin entrapment, etc
* Electronic gastroscopy is to be performed
* Voluntary informed consent

Exclusion Criteria:

Absolute contraindications:

* Patients without surgical conditions or refusing any abdominal surgery (once the capsule is stranded, it cannot be removed by surgery)
* There is a pacemaker in the body, except that the pacemaker is a new MRI compatible product
* Electronic devices such as cochlear implants, magnetic metal drug infusion pumps, nerve stimulators and magnetic metal foreign bodies are implanted in the body;
* .Women during pregnancy

Relative contraindication:

* Gastrointestinal obstruction, stenosis, and fistula are known or suspected
* Dysphagia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluating the clinical usefulness of MCE in assessing the efficacy of gastro-oesophageal varices treated under gastroscopy. | 15-30 minutes
  Comparing the value of MCE and gastroscopy in the grading of esophagogastric varices

CONTACTS AND LOCATIONS:
Overall Officials: Duowu Zou, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] European Association for the Study of the Liver. EASL Clinical Practice Guidelines for the management of patients with decompensated cirrhosis. J Hepatol. 2018 Aug;69(2):406-460. doi: 10.1016/j.jhep.2018.03.024. Epub 2018 Apr 10. No abstract available. PMID 29653741
- [Result] Cremers I, Ribeiro S. Management of variceal and nonvariceal upper gastrointestinal bleeding in patients with cirrhosis. Therap Adv Gastroenterol. 2014 Sep;7(5):206-16. doi: 10.1177/1756283X14538688. PMID 25177367
- [Result] de Franchis R; Baveno VI Faculty. Expanding consensus in portal hypertension: Report of the Baveno VI Consensus Workshop: Stratifying risk and individualizing care for portal hypertension. J Hepatol. 2015 Sep;63(3):743-52. doi: 10.1016/j.jhep.2015.05.022. Epub 2015 Jun 3. No abstract available. PMID 26047908
- [Result] Garcia-Tsao G, Abraldes JG, Berzigotti A, Bosch J. Portal hypertensive bleeding in cirrhosis: Risk stratification, diagnosis, and management: 2016 practice guidance by the American Association for the study of liver diseases. Hepatology. 2017 Jan;65(1):310-335. doi: 10.1002/hep.28906. Epub 2016 Dec 1. No abstract available. PMID 27786365
- [Result] Groszmann RJ, Garcia-Tsao G, Bosch J, Grace ND, Burroughs AK, Planas R, Escorsell A, Garcia-Pagan JC, Patch D, Matloff DS, Gao H, Makuch R; Portal Hypertension Collaborative Group. Beta-blockers to prevent gastroesophageal varices in patients with cirrhosis. N Engl J Med. 2005 Nov 24;353(21):2254-61. doi: 10.1056/NEJMoa044456. PMID 16306522
- [Result] Merli M, Nicolini G, Angeloni S, Rinaldi V, De Santis A, Merkel C, Attili AF, Riggio O. Incidence and natural history of small esophageal varices in cirrhotic patients. J Hepatol. 2003 Mar;38(3):266-72. doi: 10.1016/s0168-8278(02)00420-8. PMID 12586291